CLINICAL TRIAL: NCT02818413
Title: TRMC-Bio "Molecular Profiling of Gut Microbiome, Microbiome Metabolome, Serum Chemistry, and Metabolism-Associated SNPs in Elite Athletes"
Brief Title: Stool Microbiome, Pathogens, and Infectious Agents Among Olympic and Elite Athletes
Acronym: TRMC-Bio
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Thorne HealthTech, Inc (Industry)
Responsible Party: Principal Investigator, Brent A. Bauer, Professor of Medicine, General Internal Medicine, Mayo Clinic
Other Study IDs: 16-001515
Record Dates: First submitted 2016-06-28; First posted 2016-06-29 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Athletic Performance
Keywords: Stool microbiome; Stool metabolome; Single nucleotide polymorphisms
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples will be retained for future research
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- U.S. Olympic Team and elite athletes: Biospecimens will be collected from and questionnaires will be administered to U.S. Olympic team members and other elite athletes
  Interventions: Other: Biospecimen collection and questionnaires

INTERVENTIONS:
Other: Biospecimen collection and questionnaires — Biospecimen collection and questionnaires

SUMMARY:
This research is being done to investigate fecal microbiome and metabolome as well as serum analytes and single nucleotide polymorphisms in Olympic athletes in comparison with other elite athletes.

DETAILED DESCRIPTION:
Olympic athletes, non-Olympic elite athletes, and other active adults may have genetic and metabolic profiles that are unique. These profiles may contribute to the caliber of their athletic performance, and they may provide keys to understanding select genetic and metabolic conditions.

Therefore, the specific aims of this project are as follows:

* Specific Aim 1: Characterize the fecal microbial communities in athletes participating in the summer 2016 games and in athletes not participating in the Olympic games
* Specific Aim 2: Characterize the fecal microbiome metabolome (untargeted) in athletes participating in the summer 2016 games and in athletes not participating in the Olympic games
* Specific Aim 3: Characterize selected serum analytes and single nucleotide polymorphisms (SNPs) of elite athletes participating in the Summer 2016 games and in athletes not participating in the Olympic games, via serum and saliva analyses, respectively
* Specific Aim 4: Retain specimens from Olympic athletes participating in the summer 2016 games and in athletes not participating in the Olympic games for future research
* Specific Aim 7: Examine for the presence of Zika virus RNA in study participants who exhibit symptoms

Stool, urine, and blood specimens will be collected to study the stool metabolome, as well as serum analytes and single nucleotide polymorphisms, and the nature and extent of exposure to pathogens and infectious agents. These will be compared between Olympic athletes and other non-Olympic elite athletes.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Summer 2016 U.S. Olympic team and/or other elite athlete
* English speaking
* Willing to provide informed consent and biospecimens
* Willing to complete questionnaires regarding normal bowel habits and general health

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the U.S. Olympic teams and other elite athletes
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Baseline identification of microbial community present in stool | Approximately 1 week after collection of stool sample

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Bauer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No